CLINICAL TRIAL: NCT02388971
Title: A Randomized, Double-Blind Placebo- Controlled Phase 2a Study to Assess the Effect of CCR2 Antagonism by MLN1202 on Atherosclerotic Inflammation in Subjects With Stable Atherosclerotic Cardiovascular Disease Using FDG PET/CT Imaging
Brief Title: Proof of Mechanism Study of MLN1202 on Atherosclerotic Inflammation in Participants With Stable Atherosclerotic Cardiovascular Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study has withdrawn.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MLN1202-2006; U1111-1159-5742 (Registry Identifier: WHO)
Record Dates: First submitted 2015-02-23; First posted 2015-03-17 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: Drug therapy
MeSH Terms: conditions — Atherosclerosis | interventions — plozalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MLN1202 Dose (Experimental): MLN1202 Dose, intravenously (IV), once on Days 1, 29 and 57.
  Interventions: Drug: MLN1202
- MLN1202 Placebo (Experimental): MLN1202 placebo, intravenously (IV), once on Days 1, 29 and 57.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MLN1202 — MLN1202 solution
  Arms: MLN1202 Dose
Drug: Placebo — MLN1202 placebo-matching solution
  Arms: MLN1202 Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of MLN1202 on arterial inflammation in participants with stable atherosclerotic cardiovascular disease (CVD) who are receiving standard-of-care (SOC) therapy.

DETAILED DESCRIPTION:
The drug being tested in this study is called MLN1202. MLN1202 is being tested to treat people who have stable atherosclerotic cardiovascular disease (CVD). This study will look at changes in arterial inflammation in people who take MLN1202 in addition to standard-of-care (SOC) therapy.

The study will enroll approximately 108 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* MLN1202 Dose A intravenously (IV)
* Placebo (dummy inactive solution) - this is a solution that looks like the study drug but has no active ingredient

All participants will receive IV administration of MLN1202 or placebo on Day 1, Day 29, and Day 57 of this study.

This multi-centre trial will be conducted in the United States. The overall time to participate in this study is 19 weeks. Participants will make 7 visits to the clinic, and will be contacted by telephone approximately 35 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form (including consent for pharmacogenomics [PGx] collection) and any required privacy authorization prior to the initiation of any study procedures.
2. Is male or female and aged 35 to 80 years, inclusive at Screening.
3. Has documented atherosclerotic vascular disease (eg, coronary artery disease (CAD), peripheral arterial disease, aortic atherosclerosis or abdominal aortic aneurysm (<5 cm), carotid disease, or cerebrovascular disease) and has been clinically stable for at least 3 months prior to Screening. Documentation sufficient to demonstrate presence of atherosclerotic vascular disease will include one or more of the following:

   * i. History of myocardial infarction.
   * ii. History of stroke.
   * iii. Framingham score indicating >20% 10-year risk in an individual who is age >55.
   * iv. Documentation of atherosclerotic disease by objective diagnostic testing.
4. Are willing to undergo 2, 2-deoxy-2-[^18F]-fluoro-D-g1ucose positron emission tomography (FDG PET)/CT scans, have a body weight compatible with their imaging center's PET/CT scanner table limits and be able to tolerate the imaging procedure.
5. Are statin naïve or are taking a stable statin dose AND, if taking a statin, are not on a high dose of a high-potency statin. A high-dose of high potency statin is defined as atorvastatin ≥40 mg/day or rosuvastatin ≥20 mg/day. Furthermore, statin dose must be stable for at least 6 weeks prior to Screening FDG PET /CT scan and must not be changed during the remainder of the study.

Exclusion Criteria:

1. Has a history or clinical manifestations of:

   * a) Type 1 diabetes mellitus.
   * b) Significant heart failure (eg, New York Heart Association class III or IV).
   * c) Active or chronic liver disease.
   * d) Any chronic systemic inflammatory condition requiring ongoing therapy with anti-inflammatory drugs.
   * e) Any history of cancer, except basal cell carcinoma which has been in remission for at least 5 years prior to Day 1 of this study.
   * f) Any infection requiring antibiotic therapy within 6 weeks prior to Screening FDG PET/CT.
   * g) Any acute infection within 2 weeks of Screening FDG PET/CT scan.
   * h) Impaired renal function (estimated creatinine clearance <60 ml/min as calculated by the Cockcroft Gault formula). Re-testing may be allowed on a case by case basis.
2. Requires ongoing therapy with any systemic anti-inflammatory drugs (except nonsteroidal anti-inflammatory drug [NSAIDs]), including systemic anti-inflammatory steroids, methotrexate, colchicine, anti-inflammatory biologics, or any other compound that in the opinion of the investigator has a substantial anti-inflammatory effect.
3. Has received treatment with systemic immunosuppressant or systemic anti- inflammatory medications within 6 weeks prior to Screening FDG PET/CT scan.
4. Has a history of hypersensitivity or allergies to any component of the study medication or history of hypersensitivity to monoclonal antibodies.
5. Has any significant medical condition(s) which, in the investigator's opinion, may interfere with the participant's optimal participation in the study.
6. Has poorly controlled blood glucose, defined for the purposes of this study as glycosylated hemoglobin (HbA1c) ≥7.75% at Screening.
7. Screening FDG PET/CT scan has inadequate vascular uptake (target to background ratio [TBR] <1.6) in all of the index vessels (ascending aorta, left carotid, right carotid) as assessed by the imaging core laboratory.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
The change in arterial FDG uptake from MLN1202 treatment relative to placebo, comparing pretreatment and 3 month post-treatment time points | Baseline and 3 month post-treatment
  The primary imaging endpoint of interest is the FDG uptake, measured as a target to background ratio (TBR) within the most diseased segment (MDS) of the index vessel.

SECONDARY OUTCOMES:
The change in arterial FDG uptake from MLN1202 treatment relative to placebo, comparing pretreatment and 3 month post-treatment time points in subjects identified using a dominant model of the snip in the MCP-1 polymorphisms [MCP-1 -2518 (rs1024611)]. | Baseline and 3 month post-treatment
Change from Baseline in Mean Carotid Vessel MDS TBR | Baseline and Day 82
  Average mean of the maximum TBR in the MDS of the combined right and left carotid artery walls will be measured using 2-deoxy-2-[18F]-fluoro-D-g1ucose positron emission tomography/computed tomography (FDG PET/CT).
Change from Baseline in Mean Active Segment TBR | Baseline and Day 82
  TBR will be measured in both ascending aorta and carotids with demonstrable inflammation at Baseline using FDG PET/CT.
Change from Baseline in Mean Index Vessel TBR | Baseline and Day 82
  FDG uptake in the artery wall within the entire index vessel will be measured using FDG PET/CT.
Change from Baseline in Mean Carotid Vessel TBR | Baseline and Day 82
  The average mean of the maximum TBR and the MDS of the combined right and left carotid artery walls will be measured using FDG PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda